CLINICAL TRIAL: NCT02350829
Title: Quantification of Diffuse Myocardial Fibrosis in Children With Cardiomyopathy or Congenital Heart Disease by T1 Mapping Cardiac Magnetic Resonance
Brief Title: T1 Mapping of Diffuse Myocardial Fibrosis in Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lars Grosse-Wortmann, Cardiologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000039963
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cardiomyopathy (Active Comparator): Clinically established diagnosis of dilated, hypertrophic or arrhythmogenic right ventricular cardiomyopathy
  Adding T1 mapping sequence to the clinical cardiac magnetic resonance scan Administering Multihance 0.2ml/kg as part of clinical scan Obtaining bloodwork for assessment of hematocrit and collagen biomarkers
  Interventions: Other: Cardiac magnetic resonance sequence T1 mapping
- Congenital Heart Disease (Active Comparator): Diagnosis of Transposition of the great arteries after arterial switch operation, repaired Tetralogy of Fallot, patients after single ventricle palliation at the Fontan stage, native and repaired Aortic Coarctation Adding T1 mapping sequence to the clinical cardiac magnetic resonance scan Administering Multihance 0.2ml/kg as part of clinical scan
  Obtaining bloodwork for assessment of hematocrit and collagen biomarkers
  Interventions: Other: Cardiac magnetic resonance sequence T1 mapping
- Controls (Active Comparator): Patients undergoing a non-cardiac MR investigation (musculoskeletal / abdomen / brain) without a history of cardiac disease Adding limited cardiac sequence to the clinical magnetic resonance scan including T1 mapping Administering Multihance 0.2ml/kg as part of clinical scan Obtaining bloodwork for assessment of hematocrit and collagen biomarkers
  Interventions: Other: Cardiac magnetic resonance sequence T1 mapping

INTERVENTIONS:
Other: Cardiac magnetic resonance sequence T1 mapping — Adding T1 mapping sequence to the clinical cardiac magnetic resonance scan Obtaining bloodwork for assessment of hematocrit and collagen biomarkers

SUMMARY:
Diffuse fibrosis (or scarring) of the heart muscle is found in a variety of congenital heart diseases and in cardiomyopathies (heart muscle disease), and is considered a mediator of decreased cardiac function. The detection and quantification of diffuse myocardial fibrosis has recently become feasible non-invasively, using cardiac magnetic resonance (CMR), applying a new technique labeled T1 mapping. With this technique, the part of the heart tissue which is not made up of muscle cells (extracellular volume) can be quantified, as long as the individual's hematocrit (cellular volume in the blood) is known. The extracellular volume in the heart tissue is regarded as a quantifiable marker for the extent of diffuse myocardial fibrosis.

In the proposed study this new T1 mapping technique shall be applied in patients with different forms of congenital heart disease (n=130), cardiomyopathies (n=40) and in control subjects (n=30). The additional scan time due to participation in the study will be approximately 5-10 minutes, without changing the clinical protocol.

The main objective is to study the presence and extent of myocardial fibrosis by T1 mapping CMR in pediatric patients with congenital heart disease and cardiomyopathies, in comparison to cardiovascularly healthy controls.

DETAILED DESCRIPTION:
A better understanding of the mechanisms by which the heart muscle fails in pediatric heart disease may result in novel therapies directed at preventing rather than treating ventricular failure. The most likely mediator candidate for cardiac demise in congenital heart disease as well as the cardiomyopathies is diffuse myocardial fibrosis and non-favorable chronic biventricular remodeling. As such, fibrosis may be a marker, if not a mediator, preceding the onset of actual echocardiographic and clinical deterioration, opening opportunities for more timely and targeted treatment. Chronic stressors of myocardial function (hypoxemia, abnormal afterload or preload) appear to promote fibrosis. In some groups of patients, a genetically upregulated collagen metabolism seems to play a role. In adult patients with dilated cardiomyopathy the extent of myocardial fibrosis is predictive of outcome.

With cardiac magnetic resonance imaging, the characterization of myocardial tissue is possible. Whereas standard late gadolinium enhancement (LGE) CMR can only identify patchy scars neighboring healthy tissue, quantification of diffuse myocardial fibrosis in the living has become feasible with the T1 mapping technique. Both techniques (T1 mapping and LGE) are based on the principle that MR contrast medium (gadolinium) is trapped in between collagen fibres and is retained in areas of fibrosis while it is quickly washed out of healthy myocardium. As gadolinium is a T1 shortening agent, the fibrosed tissue with its 'trapped' gadolinium has a shorter T1 time than healthy tissue. T1 mapping measures the T1 time constant, which has been shown to correlate with the degree of fibrosis. In a refined approach of this technique, which we will use, it is now possible to quantify the extracellular space (equivalent to the degree of fibrosis) by T1 mapping. This method has been validated against the current gold standard of surgical myocardial biopsy.

ELIGIBILITY:
Inclusion Criteria: Patients with cardiomyopathies (clinically established diagnosis of dilated or hypertrophic cardiomyopathy) / Patients with congenital heart disease (Diagnosis of Transposition of the great arteries after arterial switch operation, repaired Tetralogy of Fallot, patients after single ventricle palliation at the Fontan stage) scheduled for an MR investigation including gadolinium (MRI contrast medium)

* Patients / guardians capable of giving informed consent
* Informed written consent / assent by the parents / legal guardians and patients where applicable
* Ability to undergo a MRI examination without anaesthesia. Children > 6 years are typically able to cooperate sufficiently.
* Control Patients: Patients undergoing a non-cardiac MR investigation (musculoskeletal / abdomen / brain) including gadolinium without a history of cardiac disease

Exclusion Criteria:- Consent / assent refusal by guardian / patient

* General contraindications for a MRI examination such as non-MRI compatible metallic implants, claustrophobia.
* No contrast required for the clinical portion of the MRI
* Patients who require anaesthesia for MRI (typically < 6 years of age)
* Known renal failure or previous allergic reaction to gadolinium containing contrast agent
* Control subjects: history of cardiac problems, e.g. rhythm disorders, former myocarditis, active myositis or other inflammatory conditions except suspected or confirmed inflammatory bowel disease such as Crohn's disease or ulcerative colitis
* Known pregnancy or breast feeding

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2014-02; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Measuring degree of diffuse myocardial fibrosis | Once at the end of the visit
  Participants will be followed for the duration of hospital visit, which is approximately 2 hours for the MRI part, and eventually longer, depending on possible other appointments on that day

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grosse-Wortmann, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada